CLINICAL TRIAL: NCT04161508
Title: Enhanced Recovery After Surgery in Elderly Patients: Effects of Sugammadex on Recovery After Anterior Cervical Spine Surgery
Brief Title: Enhanced Recovery After Surgery for Anterior Cervcial Spine Surgeries in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Ya-Chun Chu, MD, PhD, Chief of Division of Neuroanesthesia, department of Anesthesiology, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-06-003B
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Other Fusion of Spine, Cervical Region
Keywords: sugammadex, anterior cervical spine surgery
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated into one of the two group: neostigmine and sugammadex group for reversal of neuromuscular blockade
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization and drug preparation are executed by a nurse anesthetist according to the body weight of the patients. The nurse anesthetist is not responsible for perioperative anesthetic care, and outcome assessemnt. The volume of drugs is adjusted to 10 ml with addition of normal saline to become undifferent in appearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex (Experimental): sugammadex 2 mg/ Kg for the reversal of neuromuscular blockade at the end of surgery
  Interventions: Drug: Sugammadex Injection
- Neostigmine (Active Comparator): neostigmine 50 mcg/Kg + glycopyrrolate 10 mcg/kg for the reversal of neuromuscular blockade at the end of surgery
  Interventions: Drug: Neostigmine Injection

INTERVENTIONS:
Drug: Sugammadex Injection — injection of sugammadex for the reversal of neuromuscular blockade at the end of the surgery
  Arms: Sugammadex
Drug: Neostigmine Injection — injection of neostigmine for the reversal of neuromuscular blockade at the end of the surgery
  Other Names: glycopyrrolate
  Arms: Neostigmine

SUMMARY:
Elderly patients are subjected to airway and other complications after cervical spine surgeries. The study aim to investigate the efficacy of sugammadex (vs. neostigmine) in the recovery after anterior cervical spine surgery.

DETAILED DESCRIPTION:
Cervical spine surgeries have been increasing for many years. In Taiwan, according to the data published by the Department of Statistics, Ministry of the Interior, the elderly population (≥ 65 years old) increased and comprised 14.4% of the whole population in March, 2018. The percentages is likely to rise to 20% after 8 years. Because cervical spine surgery is a procedure commonly performed in elderly patients, the increasing trend of cervical spine surgery will likely continue. Elderly patients experienced an increased odds of length of stay ≥ 5 days, pulmonary complications, cardiac compilations, venous thromboembolism, UTI, sepsis, and unplanned readmission after anterior cervical spine surgeries according to the literature. For example, in patients ≥ 65 years old undergoing cervical spine surgery, 9.80% patients experienced at least 1 complication or death. Patients of 70~74 years old (odds ratio [OR] =1.94, 95% confidence interval [CI] = 1.03~3.65) and patients with at least 1 postoperative complication (OR 9.59, 95% CI 5.17~17.80) had increased risks of unplanned readmissions. Patients ≥ 75 years old were at higher risk of developing a complication or death with an odds ratio (OR 1.72, 95% CI 1.13~2.61). Identification of factors and change the policy of standard care in elderly patients can improve surgical outcome. The elderly have a different physiological change, such as lower elimination of the anesthetics, resulting in the confusion or delaying of detecting complications after the surgery.

Airway complications after ACCS are not uncommon. This includes sorethroat, vocal cord paresis without overt symptoms, vocal cord palsy or dysphonia, and dysphagia. The incidence of voice and swallowing complaints is primarily published in the spine literature and is inconsistent with rates ranging between 0.4% and 71%. The discrepancy may result from differences in the measurements and timepoints. We have performed a preliminary observational study investigating postoperative dysphonia and dysphagia after anterior cervical spine surgeries. We demonstrated more patients score none or mild dysphonia after surgeries in groups receiving sugammadex as a reversal of muscle relaxants. Suggammadex is a unique neuromuscular reversal drug; modified γ-cyclodextrin that allows binding encapsulation of rocuronium. The rocuronium molecule (a modified steroid) bound within sugammadex's lipophilic core, is rendered unavailable to bind to the acetylcholine receptor at the neuromuscular junction and results in the revesal of the effect of neuromuscular blackade. As the preliminary observation was not a randomized, blinded study, whether sugammadex posses beneficial effect on postoerative dysphonia warrants investigation.

Enhanced Recovery After Surgery (ERAS) proposes a multimodal, evidence-based approach to perioperative care. The first goal of ERAS is the improvement of surgical outcomes and patient experience, with a final impact on a reduction in the hospital length of stay (LOS). The implementation of ERAS in spinal surgery is in the early stages. We believe the elements for ERAS should direct to the specific characteristics of surgery and surgical population. Therefore, our investigation for improving posteropative dyshonia and dysphagia will provide a important reference for choice of elements for ERAS of cervical spine surgeries in the future.

ELIGIBILITY:
Inclusion Criteria:

anterior cervical spine surgery American society of anesthesiologist (ASA) physical status I~III

Exclusion Criteria:

unstable cervical spine requiring immobilization orthosis previous allgery to rocurium, sugammadex, and neostigmine anticipated difficult tracheal intubation preoperative sorethroat, dysphoina or dysphagia history, regardless of etiology lack of informed consent

-

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-20 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
mean time to 90% TOF ratio | up to postoperative 2 hour
  time from injection of drug to train of four ratio to 90%
mean time to extubation | up to postoperative 3 day
  time from injection of drug to tracheal extubation

SECONDARY OUTCOMES:
postoperative sorethroat | postoperative Day 1, 2,3,7,10,30
  verbal numerical rating scale (0~10, 0 denotes no sorethroat; 10 denotes maximal sorethroat)
postoperative dysphonia | postoperative Day 1, 2,3,7,10,30
  subjective assessment of voice change in horaseness, pitch, and loudness(0, 1, 2; 0 denotes none or no change; 1 denotes mild change; 2 denotes obvious change)
postoperative dysphagia | postoperative Day 1, 2,3,7,10,30
  subjective assessment of dsyphagia by Bazaz classification (based on the easiness to swallow liquid or solid food, the severity is classified into none, mild, moderate and severe)

OTHER OUTCOMES:
postoperative muscle power | postoperative 2 hour, Day 1
  the grading of muscle power (MRC):0~5, 0 denotes complete paralysis, 5 denote normal power
time to left off bed | up to postoperative 14 day
  time to patient can left off from bed
time to remove foley catheter | up to postoperative 7 day
  time to the foley catheter can be removed from patient
complications | up to postoperative 14 day
  any occurrence of global, respiratory and cardiovascular adverse events
hospital day | up to postoperative 14 day
  total day that patients are kept in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Chun Chu, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan